CLINICAL TRIAL: NCT02329249
Title: Pharmacological Aids for Interactive Smoking Cessation
Acronym: NRT_2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Center for Applied Science, Inc. (Industry)
Responsible Party: Principal Investigator, Susan Schroeder, Research Scientist, Oregon Center for Applied Science, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBIR37R-2; R44CA077986 (NIH)
Record Dates: First submitted 2014-12-29; First posted 2014-12-31 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; coach-supported; tobacco use cessation; online; internet-based; tailored
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smokefree Partners: 21 Days to Freedom (Experimental): Smoking cessation website program with live personal coach
  Interventions: Behavioral: Smokefree Partners: 21 Days to Freedom
- Wait-list control (Other): 120-day wait-list and then provided access to the smoking cessation website
  Interventions: Other: Wait-List Control

INTERVENTIONS:
Behavioral: Smokefree Partners: 21 Days to Freedom — Treatment subjects, who chose a quit date, were given 21 sessions to be viewed one session (i..e, one day) at a time, and an in-person smoking cessation coach to support them through their quit process via tailored email or phone coaching messages. Treatment users were encouraged to use pharmacological aids in their quit attempt, but smoking cessation aids were not provided.
  Other Names: Pharmacological Aids for Interactive Smoking Cessation
  Arms: Smokefree Partners: 21 Days to Freedom
Other: Wait-List Control — Subjects randomized to the control condition were placed on a wait-list and given access to the smoking cessation program after 120 days and completion of the 120-day follow-up assessment.
  Arms: Wait-list control

SUMMARY:
There is an important need for effective smoking cessation programs that both (a) promote the effective use of pharmacological aids, such as nicotine replacement products and bupropion, and (b) provide cognitive-behavioral support for stopping smoking.The Internet is an increasingly attractive intervention medium for delivering behavior change interventions, including smoking cessation.This study examined smoking cessation rates among adults participating in a randomized controlled trial of the Smokefree Partners: 21 Days to Freedom ™ program, a theoretically based, online smoking cessation program that included message tailoring and interactivity combined with the live personal support of a smoking cessation coach. Coaching support was provided almost entirely asynchronously via prescripted but individually tailored emails.

DETAILED DESCRIPTION:
The Smokefree Partners: 21 Days to Freedom combined online video, text, and interactive tools to promote the effective use of pharmacological aids (PA) - nicotine replacement products and bupropion (Zyban®) - and provide cognitive-behavioral support for users as they attempted to stop smoking. Smoking cessation content was based on the U.S. Surgeon General's Clinical Guidelines, Treating Tobacco Use and Dependence, 2008 update. Presentation of some of the content (e.g., gender of the narrator, PA recommendations) was tailored to the user on demographic and smoking history information provided during registration and within the introductory session.

Two critical features provided social support and accountability. First, each user was assigned a "live" smoking cessation coach to provide support via individually tailored phone or email contacts (contact preference specified by the user). Users also received automated email reminders and prompts from the program. Second, a bulletin board/forum feature was added to promote social support among users.

The Smokefree Partners intervention was a multi-session intervention in which users experienced a controlled and scheduled exposure to 21 discrete web site sessions. The program required users to wait at least 10 hours between sessions (i.e., login was "locked" until 10 hours had passed after a user's previous Web site session). Carefully timed and tailored coaching messages provided cessation tips and prompted users to return to the web site to view the next session.

The program was evaluated online in a randomized clinical trial of smokers recruited through major worksites across the United States. The aim of the evaluation was to determine if a theoretically based, online smoking cessation program that included message tailoring and interactivity combined with the live personal support of a coach would result in improved quit rates when compared to a wait-list control condition.

ELIGIBILITY:
Inclusion Criteria:

* large worksites with internet connection
* thinking of quitting smoking
* 18 years of age or older

Exclusion Criteria:

* not thinking of quitting smoking
* 17 years of age or younger

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2001-02; Primary Completion 2005-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Smoking cessation | 120 days
  Current smoking status was determined with two items: (a) a stage of change measure indicating smoking status and (b) a measure indicating the number of cigarettes smoked in the past 7 days. Abstinence at 30-day posttest and 120-day follow-up was confirmed by the participant choosing both (a) the response of "I do not currently smoke; I quit in the last 6 months" to the stage of change measure and (b) a response of "0" to the question "During the past 7 days, how many cigarettes did you smoke each day?"

SECONDARY OUTCOMES:
Intentions to quit smoking | 30 days and 120 days after baseline
  1 item assessing the user's likelihood of quitting smoking within the next 30 days; 1-5 response scale (1=extremely likely, 5=not at all likely)
intentions to quit and remain smokefree | 30 days and 120 days after baseline
  1 item assessing the likelihood of quitting and remaining smokefree; 1-5 response scale (1=extremely likely, 5=not at all likely)
self-efficacy for quitting | 30 days and 120 days after baseline
  2 items assessing the user's confidence to (a) quit smoking and (b) quit and remain smokefree; 1-5 response scale (1=extremely confident, 5=not at all confident)
intentions to use a pharmacological smoking cessation aid (PA) | 30 days and 120 days after baseline
  2 items assessing the user's intention to use (a) a nicotine replacement product or (b) Zyban during this quit attempt; 1-5 response scale (1=extremely likely, 5=not at all likely)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Schroeder, MPH, MCHES, Principal Investigator — Oregon Center for Applied Science